CLINICAL TRIAL: NCT07367659
Title: Comparison of the Effectiveness of Different Non-Pharmacological Methods in Reducing Injection Pain in Preschool Children: Randomized Controlled Trial
Brief Title: Non-Pharmacological Methods in Reducing Injection Pain
Acronym: Randomized
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, öznur tiryaki, Associate Professor, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: TiryakiÖ.
Record Dates: First submitted 2026-01-17; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Pain; Preschool Age Children; Injection; Fear
MeSH Terms: conditions — Pain | interventions — PALM protein, human

STUDY DESIGN:
Intervention Model Description: 32 intervention, 1 control
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- intervention group Palm (Experimental): Palm stimulator
  Interventions: Other: Palm
- intervention group ShotBloker (Experimental): ShotBloker device
  Interventions: Other: ShotBlocker
- intervention group HSTT (Experimental): HSTT application
  Interventions: Other: HSTT
- Control group (No Intervention): Rutin

INTERVENTIONS:
Other: ShotBlocker — ShotBlocker is a flat, horseshoe-shaped device used to reduce pain during subcutaneous or intramuscular (IM) injections. It features short, blunt, non-sharp projections approximately 2 mm in height and is designed to be placed against the skin, with a central opening that exposes the injection site. The device is applied to the skin just prior to injection, with its textured surface making contact with the skin. Although the projections do not penetrate the skin, they are believed to create a sensory stimulus associated with pain modulation based on the gate control theory.
  Arms: intervention group ShotBloker
Other: HSTT — Helfer Skin Tap Technique: After determining the injection site, gently tap the skin several times with the fingertips of the dominant (most commonly used) hand for approximately 5 seconds to relax the muscle. After the skin is wiped with antiseptic solution and stretched, the cap of the syringe in the dominant (most commonly used) hand is opened. A large V is made with the thumb and index finger of the non-dominant hand. The skin is tapped three times quickly using the whole hand to stimulate the major muscle fibers. The nurse/midwife counts to 3, and the needle is inserted into the muscle at a 90-degree angle simultaneously. To remove the needle from the skin, the skin is tapped three times quickly (again in a V shape) with the whole non-dominant hand, and the needle is withdrawn simultaneously with the final tap (tapping).
  Arms: intervention group HSTT
Other: Palm — The Palm Stimulator is 1.6 cm in diameter and 4 cm in length, and has a cylindrical, non-slip, and easy-to-grip structure designed to maximize palm contact. The Palm Stimulator is used by gripping it in the palm during injection. The device has blunt protrusions all around the palm to provide tactile stimulation. These blunt protrusions do not penetrate the skin but, according to gate control theory, create stimulation and close the pain gate in the spinal cord, reducing the pain perceived during injection. The researcher will show the Palm Stimulator, the device providing tactile stimulation, and allow examination. Twenty seconds before the injection, the Palm Stimulator will be placed in the palm of the child's dominant hand so that the child can grasp it. The child will be instructed to hold the device firmly in their palm throughout the procedure. After the injection is complete, the device will be removed from the child.
  Arms: intervention group Palm

SUMMARY:
In emergency departments, various methods can be used to reduce the pain experienced by children. However, the most important requirement is that the selected method provides rapid and effective results. Accordingly, it is essential that interventions performed in emergency settings are carried out in a way that enables children to experience the least possible pain and anxiety and that the long-term effects of pain are prevented. Recently, the Helfer Skin Tap Technique (HSTT), which is applied to reduce stress and pain, and the palm stimulator, which is held in the palm and has raised projections on its surface to reduce pain perception by facilitating distraction, have attracted attention. ShotBlocker is a noninvasive, U-shaped plastic device with small projections that is used to reduce injection-related pain in children who are sensitive to pain. In addition, a bee-shaped device called Buzzy®, which combines external cold application and vibration, is also widely used. These methods have been proven to be effective in reducing pain in pediatric patients during invasive procedures such as intramuscular injections and intravenous cannulation.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 4 and 6 years,
* An intramuscular (IM) medication order was prescribed by a physician,
* The IM injection was administered in the pediatric emergency department,
* No history of chronic pain-causing illness,
* No diagnosis of neurodevelopmental disorders,
* Had not received any analgesic medications in the past 6 hours,
* No history of syncope (fainting) during previous injections,

No diagnosis of mental retardation,

* No scar tissue or muscle atrophy at the intended injection site,
* Body mass index (BMI) percentile between the 10th and 90th percentiles for age and gender,
* Both child and parent provided informed consent to participate in the study.

Exclusion Criteria;

* Participants were excluded from the study if:
* The child was younger than 4 or older than 6 years,
* There was scar tissue or muscle atrophy at the injection site,
* The child or parent had communication difficulties,
* The child's BMI was below the 10th percentile (cachectic) or above the 90th percentile (obese),
* Either the child or parent declined to participate in the research.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2025-12-25 (Actual); Primary Completion 2026-01-15 (Actual); Study Completion 2026-01-17 (Actual)

PRIMARY OUTCOMES:
Pain Rating Scale | 6 weeks
  The Wong-Baker FACES Pain Rating Scale was used to assess self-reported pain levels. This scale consists of six facial expressions ranging from "no hurt" (0) to "hurts worst" (10), allowing children to select the face that best represents their level of pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Sakarya University, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Ethically, patient information can be shared upon reasonable request without revealing their identities for security reasons